CLINICAL TRIAL: NCT01982565
Title: A Clinical Pilot Study of an Oxides of Nitrogen Generating Gel Dressing System to Stimulate Healing in Diabetic Foot Ulcers
Brief Title: Nitric Oxide Generating Gel Dressing in Patients With Diabetic Foot Ulcers
Acronym: ProNOx1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Edixomed Ltd (Industry)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDX 110
Record Dates: First submitted 2013-10-24; First posted 2013-11-13 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Nitric oxide; Nitric oxide dressing; NOx; NOx dressing; Diabetic; Foot; Ulcers; Chronic
MeSH Terms: conditions — Diabetic Foot; Ulcer; Bronchiolitis Obliterans Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Experimental): NOx dressing applied and changed at least every 2 days for 12 weeks or until ulcer is healed.
  Interventions: Device: NOx dressing
- Control Arm (Active Comparator): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: NOx dressing — The NOx dressing should be changed at least every 2 days.
  Arms: Treatment Arm
Other: Standard of Care — The clinician/podiatrist is free to use whichever treatment they would choose to use on the patient in their current clinical practice.
  Arms: Control Arm

SUMMARY:
This is a 2 part study to assess the safety and efficacy of a nitric oxide (NOx) generating dressing on chronic diabetic foot ulcers (DFU). Nitric oxide has a range of effects on the body including vasodilation and angiogenesis. It is also a potent antimicrobial. This 140 patient, randomised, controlled clinical study will assess the ability of a simple 2 part, NOx generating dressing to increase blood flow in DFUs and to improve healing in chronic DFUs compared to standard of care.

DETAILED DESCRIPTION:
This is a clinical study of a new wound dressing for diabetic foot ulcers (DFU). The dressing consists of 2 stable layers that when placed together release Nitric Oxide. In preclinical studies NOx delivery has caused significant vasodilation, angiogenesis and demonstrated potent anti-microbial activity.

In part 1 of the study, the dressing will be applied to up to 20 DFUs for a set period and the blood flow in and around the wound will be measured before and after application of the dressing. Any adverse events will be recorded.

If an increase in blood flow is seen and the dressing is well tolerated, part 2 will begin, which is a multi-centre, 120 patient, randomised, controlled study. 60 patients with chronic DFUs will be treated with the NOx generating dressing and 60 patients will continue to receive standard of care. The efficacy and the tolerability of the dressing will be measured.

The NOx dressing will be changed at least every 2 days and the standard of care changed as in normal clinical practice.

At weekly clinical visits the diameter, area and volume of the wound will be measured. The infective status of the wound will be assessed and the inflammatory profile of the wound will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged over 18 years.
* Diagnosed with type 1 or type 2 diabetes.
* With a chronic (present for at least 6 weeks) full-thickness foot ulcer (on or below the malleoli) not penetrating to tendon, periosteum or bone, and with a cross-sectional area between 25 and 2500 mm2.
* Patients must have pedal blood flow between normal and moderately ischaemic. Measurable as a palpable pedal pulse or in the absence of a palpable pedal pulse they must have a TcPO2 of ≥30mmHg or an ABPI of between 0.5-1.00, or > 1.2. (An ABPI of >1.2 is associated with calcification rather than ischaemia. We are including patients with an ABPI >1.2 because ABPI is measured in large arteries. NOx has the ability to dilate medium to small arterioles which are less likely to be calcified.)
* With some degree of neuropathy (as commonly seen in the Diabetes Foot Clinic).
* Able to read and understand the Volunteer Information Sheet and to provide meaningful written informed consent.
* Able and willing to follow the Protocol requirements.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Any other serious disease likely to compromise the outcome of the trial
* Participation in any clinical study during the eight (8) weeks preceding the dosing period of the study
* Wound area greater than 2500 square mm;
* Patients with severe ischaemia. Measurable as absence of palpable pedal pulse and a TcPO2 of less than 30mmhg, or ABPI < 0.5 or between 1.0-1.2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measure the safety of the NOx generating dressing | Monitored at every visit until 12 weeks or ulcer is healed and at 3 month post treatment followed
  Number of participants with adverse events during the active study period and the following 3 months post treatment
Measure the efficacy of the NOx generating dressing | Measured at every patient visit until healed or 12 weeks of treatment is reached
  The time to healing of the ulcer will be measured and compared between the NOx generating dressing arm and the standard of care arm

SECONDARY OUTCOMES:
Measure changes in ulcer blood flow. | 3 months
  In Part 1 of the study, blood flow in the ulcer will be measured by laser Doppler fluximetry before and after the NOx generating dressing is applied.
Measure changes in the inflammatory/infective status of the wounds. | Samples taken at every visit until 12 weeks or the ulcer is healed
  Samples taken at every visit will be measured for microbial content and inflammatory cytokine presence and a comparison made between the 2 arms.
Measure the rate of repeat ulcers and breakdown in healing. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Tucker, PhD, Principal Investigator — St Barts, London
Locations (10):
- United Kingdom (10):
  - St James's University Hospital, Leeds, West Yorkshire
  - Ninewells Hospital, Dundee
  - Edinburgh Royal Infirmary, Edinburgh
  - Southern General Hospital, Glasgow
  - Kings College Hospital, London
  - Pennine Acute Hospitals Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Lancashire Teaching Hospitals, Preston
  - Salford Royal, Salford
  - Pinderfields General Hospital, Wakefield